CLINICAL TRIAL: NCT02580890
Title: Role of Transcranial Direct Current Stimulation (tDCS) in Patients With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-0498
Record Dates: First submitted 2015-10-19; First posted 2015-10-20 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- tDCS active (Experimental): Stimulation will be performed with the anode placed over the right DLPFC, and the cathode placed on the left DLPFC. The applied electric current will be 2mA and is going to be applied for 20 minutes. The electrodes have a size of 35cm ² each and will be covered by sponges soaked with saline. The stimulator to be used will be the "Chattanooga Ionto ISO 13485". Stimulation will be performed for 5 days, one time per day.
  Interventions: Device: tDCS active
- tDCS sham (Sham Comparator): For the sham tDCS, the same setting will be used. However, the current is going to be applied for only 30 seconds, not being able to induce effects on neuronal excitability.
  Interventions: Device: tDCS sham

INTERVENTIONS:
Device: tDCS active — Stimulation will be performed with the anode placed over the right DLPFC, and the cathode placed on the left DLPFC. The applied electric current will be 2mA and is going to be applied for 20 minutes. The electrodes have a size of 35cm ² each and will be covered by sponges soaked with saline.
  Arms: tDCS active
Device: tDCS sham — For the sham tDCS, the same setting will be used. However, the current is going to be applied for only 30 seconds, not being able to induce effects on neuronal excitability.
  Arms: tDCS sham

SUMMARY:
The purpose of this study is to determine whether transcranial direct current stimulation (tDCS) is effective in the treatment attention deficit hyperactivity disorder (ADHD).

Randomized, double-blind Controlled Clinical Trial

Subjects Adults (between 18 and 59 years of age) with ADHD who meet the inclusion criteria and who agree to participate in the study Will recruit from advertisements and clinical referrals to a PRODAH

Active tDCS Anode - right DLPFC Cathode - left DLPFC Electric current is 2mA - Current is applied for 20 min

Sham tDCS Same assembly is used Current is applied for 30 sec

Both groups 5 stimulation sessions on consecutive days

Following tools at Baseline, 1st week, 2 st week, 3st week and 4st week Adult ADHD Self-Report Scale (ASRS) SDS - Sheehan Disability Scale CGI - Clinical Global Impression

DETAILED DESCRIPTION:
Randomized, double-blind Controlled Clinical Trial

Subjects Adults (between 18 and 59 years of age) with ADHD who meet the inclusion criteria and who agree to participate in the study Will recruit from advertisements and clinical referrals to a PRODAH

Active tDCS Anode - right DLPFC Cathode - left DLPFC Electric current is 2mA - Current is applied for 20 min

Sham tDCS Same assembly is used Current is applied for 30 sec

Both groups 5 stimulation sessions on consecutive days

Following tools at Baseline, 1st week, 2 st week, 3st week and 4st week Adult ADHD Self-Report Scale (ASRS) SDS - Sheehan Disability Scale CGI - Clinical Global Impression

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 45 years
* Established diagnosis of ADHD according to DSM V through clinical interview and diagnostic criteria applied by trained physicians.
* ASRS greater than 21 in Part A or B
* Consent form signed
* Ability to read and interpret the self-applicable scales

Exclusion Criteria:

* Medication change in the last month
* The following comorbidities:

  1. Depressive episode with BDI greater than 9
  2. Anxiety Disorder with greater than 15 BAI
  3. Bipolar Disorder with depressive symptoms, manic or hypomanic in the last 6 months
  4. Schizophrenia and other psychotic disorders
  5. Autism
  6. dependence of substances
  7. Mental retardation or dementia
* Epilepsy or anticonvulsant use
* Clinically significant medical condition
* Contraindications for tDCS (metallic implants, cranioencefálica important anatomical change ...)

Exclusion criteria retrospectively: two fouls in a row dating to stimulation or three fouls in total days.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in scores obtained in ASRS scale. | Autcome measure assesments: day 1 (pre-intervention), day 5 (post-intervention), 1 and 4 weeks later (accompaniment).
  This scale is used to access symptoms improvement in ADHD patients, is a self repor scale.

SECONDARY OUTCOMES:
Change in scores obtained in CGI scale. | Autcome measure assesments: day 1 (pre-intervention), day 5 (post-intervention), 1 and 4 weeks later (accompaniment).
  This scale is used to access clinical improvement in ADHD patients,
Change in scores obtained in Sheehan disability scale | Autcome measure assesments: day 1 (pre-intervention), day 5 (post-intervention), 1 and 4 weeks later (accompaniment).

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Schestatsky, MD, PhD, Study Director — Professor of Department of Internal Medicine, UFRGS, Brazil.; Douglas T Leffa, MD student, Principal Investigator — MD student from Federal University of Rio Grande do Sul (UFRGS), Brazil.; Luis Augusto Rohde, MD, Phd, Study Director — Professor of Department of Psychiatry, UFRGS, Brazil.; Eugenio H Grevet, MD, phD, Study Director — Associate Professor of Department of Psychiatry, UFRGS, Brazil.; Carolina T Cachoeira, MD, Principal Investigator — Federal University of Rio Grande do Sul (UFRGS), Brazil
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided